CLINICAL TRIAL: NCT02266199
Title: Validation of a New Questionnaire Regarding Pain Management in Hospitals Using a Qualitative Verification
Brief Title: Validation of a New Questionnaire Regarding Pain Management
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr., Ruhr University of Bochum
Other Study IDs: VNQI-2012
Record Dates: First submitted 2013-08-22; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: questionnaire; quality assurance; qualitative Verification; conservative patients; interview
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- conservative patients: in-patients on pneumology, cardiology, neurology, gastroenterology, endocrinology
- operative patients: inpatient on Traumatology, Plastic Surgery, Cardiothoracic Surgery, Gynecology, Abdominal Surgery

SUMMARY:
The study includes operative as well as conservative patients using a questionnaire containing items of pain quality. After having completed the questionnaire, the patient is interviewed by an assistant. By this way the new questionnaire should be validated.

In addition the patient´s personal experiences are included and conservative patients can be compared to operative patients.

DETAILED DESCRIPTION:
It is validated whether the questions are formulated comprehensively and the patient consequently is able to understand all the different interrogated aspects of the questionnaire.

Exemplarily the patient is asked to express his pain in an analogue scale in various situations and which type of pain they experience (for example headache).

Moreover, it is tested whether there is a relation between the pain and the treatment he receives, and whether the patient expressed the need for additional medication.

Besides, it is asked whether he already took medication before his hospitalisation.

With help of the interview, which is conducted subsequent to the questionnaire, it is verified if the patient understands the aspects. Some of the questions are interrogated in depth by additional questions, for example which type of pain he experiences in which situation.

One important aspect is to find out whether the patient is conscious about his medication.

In order to do so, schedules are used, which are based on the documented patient's history.

ELIGIBILITY:
Inclusion Criteria:

* Signing the consent form
* Patients with acute postoperative pain
* Patients with acute pain with conservative treatment
* Patients with ≥ 18 years of age

Exclusion Criteria:

* Lack of signature of the informed consent
* All physical and mental impairments which don´t allow the completion of the questionnaire or answering the interview
* Difficulties with the German language
* <18 years of age
* Isolation of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are all conservative and postoperative patients who are inpatients on pneumology, cardiology, neurology, gastroenterology, endocrinology, Traumatology, Plastic Surgery, Cardiothoracic Surgery, Gynecology, Abdominal Surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Interview | 10-60 minutes
  directly after answering the questionnaire, the patients are interviewed face-to-face about the personal background to answer the questions that way and does they understood the questions like the experts

SECONDARY OUTCOMES:
Pain intensity | 10-60 minutes
  The pain intensity of the current pain, the exercise-related pain and the worst pain intensity in the last 24h is specified by the numerical rating scale ranging from 0-10 (NRS with 0 = no pain and 10 = worst pain imaginable)
Grading of pain management | 10-60 minutes
  using a grading scale 1 (very good) - 6 (unsufficient)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr., Study Director — Bergmannsheil Bochum
Locations (3):
- Germany (3):
  - Bergmannsheil, department for pain management, Bochum, North Rhine-Westphalia
  - Knappschaftskrankenhaus, Langendreer, North Rhine-Westphalia
  - Marienhospital, Witten, North Rhine-Westphalia